CLINICAL TRIAL: NCT06403462
Title: Comparison Between Ultrasound-guided Transversus Abdominis Plane and Transversalis Fascia Plane Block for Pediatric Patients Undergoing Alveoloplasty With Iliac Bone Graft: a Prospective Randomized Controlled Trial
Brief Title: Transversalis Fascia Plane Block for Iliac Bone Graft in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-2311-167-1488
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plane block (Active Comparator)
  Interventions: Procedure: transversus abdominis plane block
- transversalis fascial plane block (Experimental)
  Interventions: Procedure: transversalis fascial plane block

INTERVENTIONS:
Procedure: transversalis fascial plane block — ultrasound guidance transversalis fascial plane block after iliac bone graft
  Arms: transversalis fascial plane block
Procedure: transversus abdominis plane block — ultrasound guidance lateral transversus abdominis plane block after iliac bone graft
  Arms: transversus abdominis plane block

SUMMARY:
The purpose of this study is to determine which method is more effective in postoperative pain control in children undergoing iliac bone grafting for alveoloplasty under general anesthesia: ultrasound-guided transverse abdominal blockade or transversalis fascia plane block

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 years and older but under 18 undergoing iliac bone grafting for alveoloplasty

Exclusion Criteria:

* Patients with diseases that affect pain sensitivity differently from the general population (e.g., congenital insensitivity to pain with anhidrosis, complex regional pain syndrome, etc.)
* Cases where there is difficulty in expressing pain (due to cognitive or functional deficits, or limited ability to communicate)
* Unstable vital signs (heart rate, blood pressure)
* Common contraindications for Ropivacaine: 1) Patients with a history of hypersensitivity to this drug or other amide local anesthetics, 2) Patients in a state of major bleeding or shock, 3) Patients with inflammation at or around the site of administration, 4) Patients with sepsis, 5) Intravenous regional anesthesia (Bier block)
* History of allergy to opioid medications
* Severe renal impairment (Creatinine >3.0mg/dL)
* Severe liver function abnormalities (aspartate transaminase > 120 unit/L, alanine aminotransferase > 120 unit/L)
* Peripheral nervous system disorders
* Other cases deemed unsuitable by the researcher

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
total consumption of opioid (mcg/kg) | from the end of surgery up to 24 hours later
  total opioid consumption at 24 hours after the end of surgery

SECONDARY OUTCOMES:
Postoperative Pain score | at 30 minutes, 1 hour, 3 hours, 6 hours, 24 hours after the end of surgery
  Pain scores is assessed by Numerical Rating Scale, which requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Total consumption of non-opioid (mg/kg) | within 24 hours after the end of surgery
  Non-opioid analgesics usage per body weight within 24 hours after surgery
Cold sensation | at 30 minutes after the end of surgery
  Evaluation of the distribution of lost cold sensation in the skin in the recovery room (Dermatomal distribution of the loss of cold sensation using an alcohol swab at post-anesthesia care unit, assessed by a blinded assessor in the Post Anesthesia Care Unit).
The incidence of side effects of analgesic medications (percent) | within 24 hours after the end of surgery
  Analgesic-related side effects (nausea, vomiting, constipation, pruritis, dizziness, dry mouth, somnolence, etc.) within 24 hours after surgery.
Satisfaction score | at 24 hours after the end of surgery
  Patient satisfaction score (0-100 points, with 100 being very satisfied and 0 being very dissatisfied).
Sleep quality score | at 24 hours after the end of surgery
  Quality of sleep on the day of operation (satisfaction score, 0-100 points, with 100 being very satisfied and 0 being very dissatisfied).
Procedure time (min) | within 10 minutes after the end of surgery
  total procedure time from needle puncture to the end of block
First ambulation (hours) | within 24 hours after the end of surgery
  Time to first ambulation (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea